CLINICAL TRIAL: NCT06869096
Title: A Comparative Study of Chlorhexidine Versus Saline Irrigation of the Surgical Area During Colorectal Cancer Surgery: a Multicenter, Stratified Randomized Controlled Trial.
Brief Title: Chlorhexidine Gluconate Versus Saline for Flushing the Surgical Area During Colorectal Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchong Central Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024135
Record Dates: First submitted 2025-03-10; First posted 2025-03-11 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer; Surgical Site Infection; Chlorhexidine; Complications
MeSH Terms: conditions — Colorectal Neoplasms; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Diabetic rectal cancer patients, chlorhexidine irrigation group (Experimental): After colorectal cancer surgery, flush the surgical area with chlorhexidine solution 1 minute before suturing the skin.
  Interventions: Procedure: Intraoperative area irrigation
- Diabetic rectal cancer patients, saline irrigation group (No Intervention)
- Diabetic colon cancer patients, chlorhexidine irrigation group (Experimental)
  Interventions: Procedure: Intraoperative area irrigation
- Diabetic colon cancer patients, saline irrigation group (No Intervention)
- Non-diabetic rectal cancer patients, chlorhexidine irrigation group (Experimental)
  Interventions: Procedure: Intraoperative area irrigation
- Non-diabetic rectal cancer patients, saline irrigation group (No Intervention)
- Non-diabetic colon cancer patients, chlorhexidine irrigation group (Experimental)
  Interventions: Procedure: Intraoperative area irrigation
- Non-diabetic colon cancer patients, saline irrigation group (No Intervention)

INTERVENTIONS:
Procedure: Intraoperative area irrigation — After colorectal cancer surgery, flush the surgical area with chlorhexidine solution 1 minute before suturing the skin. According to abdominal cavity contamination, bleeding and tumor invasion to determine the flushing time and flush fluid volume. If the abdominal cavity infection is more serious or exudate more, the flushing time can be relatively prolonged. At last, there were no obvious blood residue, tissue fragments and suppurative secretions in abdominal cavity. Ensure that the surgical field of vision is clear, the surface of each organ is smooth, and there is no abnormal exudate.
  Arms: Diabetic colon cancer patients, chlorhexidine irrigation group; Diabetic rectal cancer patients, chlorhexidine irrigation group; Non-diabetic colon cancer patients, chlorhexidine irrigation group; Non-diabetic rectal cancer patients, chlorhexidine irrigation group

SUMMARY:
The aim of this study was to compare the effectiveness of chlorhexidine versus saline in flushing the surgical area during colorectal cancer surgery. The primary outcomes included surgical site infection, postoperative complication rates, et al.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-85 years,
2. Patients with surgically resectable colorectal tumors confirmed by CT/MRI before surgery
3. All patients had a performance status score of 0 or 1 in the Eastern Tumor Cooperative group
4. American Society of Anesthesiology grade I-III

Exclusion Criteria:

1. The tumor may have distant metastasis
2. History of previous abdominal surgery
3. The patient has a history of other malignant tumors diagnosed in the past 5 years and has received radiotherapy and chemotherapy in the past
4. There are obvious contraindications to surgery (obvious abnormal liver and kidney function, pregnancy)
5. Participated in other clinical trials within the past 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Surgical site infection within 30 days | 30 days
  Any surgical site infection within 30 days of surgery is classified as superficial incision, deep mouth, or organ space infection according to the U.S. Centers for Disease Control and Prevention standards.

SECONDARY OUTCOMES:
Number of participants with Postoperative complication within 30 days | 30 days
  Including anastomotic fistula, anastomotic hemorrhage, intestinal obstruction, deep vein thrombosis and so on

CONTACTS AND LOCATIONS:
Locations (1):
- Nanchong Central Hospital, Nanchong, Sichuan, China